CLINICAL TRIAL: NCT04887350
Title: Naturalistic Pilot Study Comparing the Feasibility of Applying a Student Senior Isolation Prevention Partnership vs. Problem-solving Therapy vs. Waitlist Control in Patients Suffering From Late-life Depression During the COVID-19 Pandemic: A Randomized Controlled Trial
Brief Title: SSIPP vs. PST vs. WLC
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Staffing shortages
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Akshya Vasudev, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11336
Record Dates: First submitted 2021-05-05; First posted 2021-05-14 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Major Depressive Disorder; Late Life Depression
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 1:1:1 ratio to one of the three study groups.
Masking Description: All study participants will be blinded to the study hypotheses to prevent expectation bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Student-Senior Isolation Prevention Partnership (SSIPP) (Experimental): The Student-Senior Isolation Prevention Partnership is a phone administered talk therapy.
  Interventions: Behavioral: Student-Senior Isolation Prevention Partnership (SSIPP)
- Problem Solving Therapy (PST) (Active Comparator): Problem Solving Therapy is a phone administered talk therapy.
  Interventions: Behavioral: Problem Solving Therapy (PST).
- Wait List Control (WLC) (Other): Participants in the WLC will continue with their regular treatments for the 12 week study period but not receive any study related intervention during this 12 weeks. Following completion of all study assessments WLC participants will self-select either SSIPP or PST. Participants in WLC will not complete study assessments after week 12.
  Interventions: Behavioral: Student-Senior Isolation Prevention Partnership (SSIPP); Behavioral: Problem Solving Therapy (PST).

INTERVENTIONS:
Behavioral: Student-Senior Isolation Prevention Partnership (SSIPP) — The Student-Senior Isolation Prevention Partnership partners medical students with older adults in the community to provide social support and connection through regular phone calls. The goal of SSIPP is to reduce rates of anxiety, depression, and loneliness, while fostering resilience among seniors in our communities. This intervention will be delivered by phone to study participants once a week for a 30-60 minute session over a 12-week period.
  Arms: Student-Senior Isolation Prevention Partnership (SSIPP); Wait List Control (WLC)
Behavioral: Problem Solving Therapy (PST). — Problem Solving Therapy is a psychotherapeutic intervention that teaches community members to identify and clarify problems at hand, set clear, achievable goals, brain-storm solutions to the problem, select their preferred solution, implement this solution, and evaluate the outcomes. This intervention will be delivered by a trained healthcare professional by phone to study participants once a week for a 30-60 minute session over a 12-week period.
  Arms: Problem Solving Therapy (PST); Wait List Control (WLC)

SUMMARY:
The COVID-19 pandemic and continued lockdown measures have led to social isolation that is likely disproportionately affecting community-dwelling seniors. This social isolation of seniors is expected to cause detrimental health effects especially in those who have an ongoing or new onset late life depressive episode. The COVID-19 pandemic has also made accessing formal psychotherapy services increasingly difficult due to an increased demand for these services and a limited number of trained professionals available to deliver these interventions. We plan to conduct an open label, pilot, randomized controlled trial (RCT), comparing a virtually delivered (telephone) student led mental health supportive initiative, Student Senior Isolation Prevention Partnership (SSIPP) (n=15) compared to a telephone delivered standard psychotherapy intervention, problem-solving therapy (PST) (n=15) versus a wait list control (n=15) in community-dwelling seniors suffering from late life depression. Participants in this study will be blinded to the hypothesis, while those performing data analysis will be blinded to treatment allocation. Both SSIPP and PST will be delivered via telephone as a weekly session for 12-weeks. Feasibility measures of recruitment, retention and costs will be collected as primary outcome measures. Self-rated measures of depression, anxiety, isolation and resilience will comprise secondary exploratory outcomes. We anticipate that it will be feasible to conduct an RCT of these telephone interventions, SSIPP and PST, in socially isolated community-dwelling seniors. Data from this study will be critical to plan a subsequent confirmatory large-scale RCT. It could be that telephone delivered medical student led supportive intervention, SSIPP and/or a telephone delivered psychotherapy initiative, PST, can be feasibly applied in the current pandemic to a high-risk population, isolated seniors suffering from depression.

DETAILED DESCRIPTION:
BACKGROUND

The rapid spread of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), the virus responsible for the current coronavirus disease 2019 (COVID-19) outbreak, has led to strict social distancing and social isolation recommendations from the World Health Organization (1). As the elderly are most susceptible to critical illness and fatality due to infection with SARS-CoV-2, they have also been subjected to the most stringent social isolation guidelines in Canada as an attempt to prevent death in this population (1,2). While these public health measures are necessary to prevent the spread of SARS-CoV-2 among our vulnerable geriatric populations and to protect our over-burdened healthcare systems, social isolation has had a detrimental impact on the mental health of this population and has been deemed a mental health crisis (1,3).

The aim of this study is to assess the feasibility of delivering SSIPP in London, Canada, as compared to an active control, PST, as well as a wait list control. Such a study would also allow to collect effect size estimates on the efficacy of SSIPP on self-rated depression, anxiety, isolation and resilience among community-dwelling seniors. As SSIPP is more accessible and more readily available than PST, we aim to determine if SSIPP is as effective as the structured psychotherapy intervention PST at achieving these outcomes. Data from this study will help inform the design of a future large, multi-center RCT.

OBJECTIVES

Objective 1: To determine if it is feasible to conduct an RCT of telephone SSIPP in comparison to PST delivered to community-dwelling seniors during the current constraints imposed by COVID-19 and the need for telephone delivery of these services.

Objective 2: To determine the extent of change in self-rated depression, anxiety, isolation and resilience measures in a telephone delivered SSIPP as compared to telephone delivered PST and wait list control among community dwelling seniors.

HYPOTHESES

Hypothesis 1: It will be feasible to conduct an RCT of telephone SSIPP in comparison to telephone PST and a wait list control, under the current constraints imposed by COVID-19 and the need for telephone delivery of these services.

Hypothesis 2: It will be possible to collect effect size estimates of SSIPP compared to PST and a wait list control on symptoms of depression, anxiety, isolation and resilience in community dwelling seniors.

STUDY DESIGN

This study will be open label, randomized, controlled trial comparing 12-week telephone delivered SSIPP and PST in a total of 45 participants, randomized in a 1:1:1 ratio to one of three groups. The three study groups that participants could be randomized to, include SSIPP, PST, or a waitlist control (WLC). The WLC participants will self-select participation in either SSIPP or PST at the end of the 12-week waiting period. They will not complete study assessments following week 12. This study will plan to enroll n=45 with 15 participants randomized to each of the three groups. Participants will be asked to complete brief surveys, online in REDCap, or over the phone with a Research Assistant at weeks 0 and 12 of the study. REDCap will be used to achieve randomization and its concealment. Statistical analysts will be blinded to group allocation during data analysis.

RECRUITMENT

Participants will include community-dwelling seniors (n=45) recruited from the Division of Geriatric Psychiatry at Parkwood Institute and from the Geriatric Mental Health Program at London Health Sciences Center, both located in London, Ontario. Participants to these two programs receive referrals from family doctors serving the city of London and surrounding Middlesex County. The study will recruit via existing relationships and referrals established by the study PI and co-investigator.

STATISTICAL ANALYSIS PLAN

Primary outcome measures will be calculated using rates, percentages and costs. For exploratory purposes, the secondary outcome measures will be subject to the following analyses. A Multivariate Analysis of Variance (MANOVA) will be conducted to detect differences between the two interventions, i.e. SSIPP and PST as the independent variables and scores on GAD-7, PHQ-9, and CD-RISC-10 scale as the dependent variables. Multivariate F value (Wilks' λ or Hotelling's trace or Pillai's trace) will be used with a statistical significance set at p < 0.05. Demographic measures will be described using either calculations of means or percentage as required. As there is no consensus or current evidence recommending an appropriate sample size for feasibility studies, it is advised that feasibility study samples sizes not be attempted a priori. Pilot studies investigating the comparable psychotherapies cognitive behavioural therapy (CBT) and mindfulness-based cognitive therapy (MCBT) were able to demonstrate reductions in self-reported anxiety and depression with a sample size of n=52 and n=30, respectively. Given these effect sizes, the desired sample size is n=45. Attrition and retention rates will be calculated as feasibility measures as part of this pilot study to help inform required sample size for a future large, multi-center RCT.

IBM SPSS ® (v26) will be used for the conduction of data analysis. Contingent on final sample size, either the Kolmogorov-Smirnov or the Shapiro-Wilk test will be used to assess normality of the data. The Expectation-Maximization (EM) algorithm will be used to account for missing data. Analysis will first be carried out using an Intent to Treat (ITT) approach, followed by per protocol (PP) analyses for the participants who completed the study only. The differences in anxiety, depression, and resiliency outcomes between the groups at week 0 and week 12 will be analyzed using a repeated MANOVA test, in both ITT and PP analysis groups.

ELIGIBILITY:
Inclusion Criteria:

1. Community-dwelling senior 65 years of age or older.
2. Meeting criteria of suffering from an episode of major depression, mild to moderate, as assessed by an experienced psychiatrist (DSM 296.21, 296.22, 296.31, 296.32), with the following applicable specifiers including anxious distress, mixed features, melancholic features, atypical features and seasonal pattern
3. Willing to receive services via telephone.
4. Have sufficient hearing to converse via telephone.
5. Have an adequate understanding of written and spoken English.
6. Answer yes to the question "do you perceive that you are either lonely or isolated?"

Exclusion Criteria:

1. Pre-existing dementia or other neurodegenerative disorder as confirmed by a Montreal Cognitive Assessment (MoCA) score, telephone version, 17 or below
2. History of schizophrenia
3. History of bipolar disorder
4. History of substance use disorder
5. History of personality disorder as per previous clinical documentation
6. History of suicide attempts or threats as per previous clinical documentation or endorsement of any of the questions from item 2-6 of the Columbia- Suicide Severity Rating Scale.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-08-09 (Actual); Primary Completion 2022-04-09 (Actual); Study Completion 2022-04-09 (Actual)

PRIMARY OUTCOMES:
Rate of participant recruitment | through study completion, an average of 1 year
  The number of participants recruited per month will be calculated by dividing the total number of participants at the end of the study by the number of study months over which recruitment took place.
Rate of retention | through study completion, an average of 1 year
  The retention rate will be calculated by dividing the total number of participants who completed a week 12 study assessment by the total number of participants enrolled in the study.
Completeness of data entry | through study completion, an average of 1 year
  Completeness of data entry will be calculated by dividing the number of completed CRF's at the end of the study by the CRF maximum potential completion number.
Cost of interventions | through study completion, an average of 1 year
  The cost of study intervention will be calculated by dividing the total number of participants who attended at least one study intervention by the total cost of interventions to determine a cost per participant.
Unexpected costs | through study completion, an average of 1 year
  Any unanticipated costs will be recorded and reported at the end of the study.

SECONDARY OUTCOMES:
Depression | Week 0, Week 12
  The Patient Health Questionnaire (PHQ-9) is a 9-item, self-rated measure of depression which has been validated for screening a major depressive episode in adults. Total scores indicate level of depression: 0-4, no depression; 5-9, mild depression; 10-14, moderate depression; 15-19, moderately severe depression; 20-27, severe depression.
Anxiety | Week 0, Week 12
  The Generalized Anxiety Disorder 7-item scale (each scored 0-3) is a self-rated measure of anxiety that has been validated for the diagnosis of Generalized Anxiety Disorder in the adult population. The scale is scored from 0 to 21. Higher scores indicate greater anxiety symptoms (5-9, mild anxiety; 10-14, moderate anxiety; 15-21 severe anxiety).
Resilience | Week 0, Week 12
  The Connor-Davidson Resilience Scale (CD-RISC) is a self-rated assessment scale comprised of 10 items, each rated on a 5-point Likert scale (0 = not true at all to 4 = true nearly all the time). Higher scores reflect greater resilience, indicating one's ability to cope with stressful situations. The scale has demonstrated strong reliability and validity in a variety of populations.
Isolation | Week 0, Week 12
  The Lubben Social Network Scale 6 is a self-rated assessment scale comprised of 6 items, each rated on a 6-point likert scale (0 = none, 1 = one, 2 = two, 3 = three or four, 4 = five thru eight, 5 = nine or more). Higher scores indicate a lower level of isolation.

CONTACTS AND LOCATIONS:
Overall Officials: Akshya Vasudev, MD, Principal Investigator — London Health Sciences Centre
Locations (1):
- London Health Sciences Centre Victoria Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Banerjee D. The impact of Covid-19 pandemic on elderly mental health. Int J Geriatr Psychiatry. 2020 Dec;35(12):1466-1467. doi: 10.1002/gps.5320. Epub 2020 Jun 27. No abstract available. PMID 32364283
- [Background] Wang L, He W, Yu X, Hu D, Bao M, Liu H, Zhou J, Jiang H. Coronavirus disease 2019 in elderly patients: Characteristics and prognostic factors based on 4-week follow-up. J Infect. 2020 Jun;80(6):639-645. doi: 10.1016/j.jinf.2020.03.019. Epub 2020 Mar 30. PMID 32240670
- [Background] Armitage R, Nellums LB. COVID-19 and the consequences of isolating the elderly. Lancet Public Health. 2020 May;5(5):e256. doi: 10.1016/S2468-2667(20)30061-X. Epub 2020 Mar 20. No abstract available. PMID 32199471

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-21): https://cdn.clinicaltrials.gov/large-docs/50/NCT04887350/Prot_SAP_000.pdf
  • Informed Consent Form (2021-07-22): https://cdn.clinicaltrials.gov/large-docs/50/NCT04887350/ICF_001.pdf